CLINICAL TRIAL: NCT05585853
Title: The Effect of Virtual Reality Glasses Applied on Chest Tube Removal After Open Heart Surgery on Pain Level and Hemodynamic Variables
Brief Title: The Effect of Virtual Reality Glasses on Pain Level and Hemo-Dynamic Variables After Open Heart Surgery
Acronym: Virtual
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Tugba CAM YANIK, Principal Investigator in the study/ Research Assistant at Surgical Nursing, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MersinUnii
Record Dates: First submitted 2022-10-12; First posted 2022-10-19 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Pain; Hemodynamic Instability
Keywords: pain; Virtual reality glasses; open heart surgery; hemodynamic
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: The study was planned as a prospective, two-armed (1:1), randomized controlled experimental study. This randomized controlled trial will be reported according to the CONSORT guidelines.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Reality application group (Experimental): Virtual reality glasses (VR Box Virtual Reality Headset 3D Vr Glasses V2.0 2020 model) compatible with the mobile phone (Lenovo P2a42) with the Android operating system will be worn and the patient will be watched (underwater world, open-air museum tours, beach trips and nature scenes) by patients for an average of 10 minutes during chest tube removal.
  Interventions: Other: virtual reality
- Standard of care (No Intervention): Only standard care will be given and no application will be made.

INTERVENTIONS:
Other: virtual reality — Virtual reality glasses application is a method without any side effects. Patients will be treated for an average of 10 minutes. Data will be collected before, during, immediately after the application, at the 15th and 30th minutes.
  Arms: Virtual Reality application group

SUMMARY:
In this study, between 1 January 2025 - 1 June 2025, who met the inclusion and exclusion criteria, a total of 82 patients who are on the 2nd or 3rd day after the surgery and who are hospitalized in the cardiovascular surgery intensive care clinic will be recruited.

DETAILED DESCRIPTION:
The patient will be put on virtual reality glasses five minutes before the chest tube is removed. Afterwards, it will continue to be watched while the tube is taken and virtual reality glasses will be watched for another five minutes. Pain level and hemodynamic variables will be checked before, during, and 15 and 30 minutes after virtual reality glasses are watched. The participants in the control group will receive routine treatment and care, and their data will be collected at the same time as those in the study group. Hemodynamic variables will be monitored and recorded on the monitor.

Virtual reality glasses application is a method without any side effects. During the research, any adverse condition (vision problem, nausea, dizziness, etc.) related to the use of virtual glasses will be observed by the researcher. Since virtual reality glasses will be used in another patient after being used on one patient, disinfection will be made in line with the company's recommendations, taking into account the pandemic conditions. Throughout the application, feedback will be received from the patients by the researchers.

ELIGIBILITY:
Inclusion Criteria:

* Agreeing to participate in the research (signing the Informed Consent Form),
* Conscious and cooperative,
* Stable hemodynamic status,
* Speaks and understands Turkish,
* Over 18 years old,
* On the 2nd and 3rd day after open heart surgery,
* Having chest tube,
* No sensitivity or trauma in the area (for the study group) where the virtual reality glasses will be applied,
* No active COVID-19 infection,
* Patients without any psychiatric diagnosis

Exclusion Criteria:

* Agreeing to participate in the research (signing the Informed Consent Form),
* Not conscious,
* Not cooperative
* Unstable hemodynamic status,
* Speaks and understands Turkish,
* who are under the age of 18,
* On the 0th or 1st day after surgery,
* No chest tube,
* Has sensitivity or trauma in the area (for the study group) where the virtual reality
* Active COVID-19 infection,
* Patients with a psychiatric diagnosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-08-26 (Actual)

PRIMARY OUTCOMES:
Pain evaluated using the Visual Analogue Scale | Change from before implementation up to 30 minutes
  Visual Analogue Scala has been developed to convert some values that cannot be measured numerically into numeric values. The VAS, which is a safe and easily applicable scale tool generally accepted in the world literature, consists of a 10 cm long line and there are subjective descriptive expressions at both ends of the scale (0 cm = none at all and 10 cm = highest degree.)

SECONDARY OUTCOMES:
Systolic blood pressure | Change from before implementation up to 30 minutes
  Systolic blood pressure (SBP), mmHg
Diastolic blood pressure | Change from before implementation up to 30 minutes
  Diastolic blood pressure (DBP), mmHg
Heart rate | Change from before implementation up to 30 minutes
  Beats per minute
Respiratory rate | Change from before implementation up to 30 minutes
  Lung breathing
Peripheral oxygen saturation | Change from before implementation up to 30 minutes
  %, percentage of oxygenated hemoglobin in peripheral arterial blood

CONTACTS AND LOCATIONS:
Overall Officials: Gülay ALTUN UĞRAŞ, PhD, Principal Investigator — Mersin University; Sevban ARSLAN, PhD, Principal Investigator — Cukurova University; Muaz GÜLŞEN, master, Principal Investigator — Cukurova University; Firdevs Ebru ÖZDEMİR, master, Principal Investigator — Mersin University
Locations (1):
- Turkey, Mersin University,, Mersin, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No